CLINICAL TRIAL: NCT04372134
Title: The Effect of High Frequency Repetetive Transcranial Magnetic Stimulation on Motor Recovery and Gait Parameters in Patients With Chronic Incomplete Spinal Cord Injury
Brief Title: The Effect of rTMS in Patients With Spinal Cord Injury (rTMS:Repetetive Transcranial Magnetic Stimulation)
Acronym: rTMS:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2020-04-08; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Spinal Cord Injury
Keywords: r TMS; spinal cord injury; motor recovery,; gait
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real rTMS group (Active Comparator): motor incomplete traumatic SCI patients receiving real repetitive transcranial magnetic stimulation therapy
  Interventions: Device: repetitive transcranial magnetic stimulation therapy
- sham r TMS (Sham Comparator): motor incomplete traumatic SCI patients receiving sham repetitive transcranial magnetic stimulation therapy
  Interventions: Device: repetitive transcranial magnetic stimulation therapy

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation therapy — A sham-controlled double-blind randomized study was undertaken. 28 patients with chronic (>1 year) motor incomplete traumatic SCI were randomized into real rTMS group (n=14) or sham rTMS group (n=14). Real rTMS (20 Hz, a total of 1600 stimuli) or sham r TMS were applied in the motor cortex area of lower extremities during 3 weeks (15 sessions). In addition to rTMS sessions, patients underwent a rehabilitation program including exercises for strengthening, walking and balance.
  Other Names: rehabilitation program

SUMMARY:
It is postulated that high frequency repetitive transcranial magnetic stimulation (rTMS) can decrease the corticospinal inhibition and enhance the motor recovery. This study is aimed to investigate the effect of high frequency rTMS on lower extremity motor recovery and gait parameters in patients with chronic motor incomplete traumatic spinal cord injury (SCI).

DETAILED DESCRIPTION:
A sham-controlled double-blind randomized study was undertaken. 28 patients with chronic (>1 year) motor incomplete traumatic SCI were randomized into real rTMS group (n=14) or sham rTMS group (n=14). Real rTMS (20 Hz, a total of 1600 stimuli) or sham r TMS were applied in the motor cortex area of lower extremities during 3 weeks (15 sessions). In addition to rTMS sessions, patients underwent a rehabilitation program including exercises for strengthening, walking and balance. Lower extremity motor score (LEMS), the temporal-spatial gait parameters measured by 3D gait analysis, Walking Index for SCI-II (WISCI-II) scale and 10 meters walking test were assessed at baseline, 3 weeks (after the treatment sessions) and 5 weeks (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis of motor incomplete cervical or thoracic spinal cord injury (ASIA C or D), spinal cord injury due to trauma at least one year previously
* the ability to walk at least 10 meters independently or with assisted devices such as cane / canadian, age (18-45 years). All participants signed the informed consent form.

Exclusion Criteria:

* the presence of other musculoskeletal or neurological diseases that may prevent walking, lower motor neuron lesion (cauda equina and conus medullaris)
* family history of epilepsy
* the presence of brain injury
* the presence of cranium defect
* the presence of pacemaker
* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
The lower extremity motor scores of the patients | through study completion, an average of 2 weeks (Change from Baseline The lower extremity motor scores of the patients at 2 weeks.)
  The lower extremity motor scores of the patients (degree of muscle strength according to the American Spinal Injury Association (ASIA) Impairment Scale )(The assesment of ASIA scale includes 5 classification as ASIA A, B,C,D,E. ASIA A is the worst score and ASIA E is the best score)

SECONDARY OUTCOMES:
the parameters of gait analysis - walking speed | through study completion, an average of 2 weeks (Change from Baseline parameters of gait analysis of the patients at 2 weeks.)
  walking speed (centimeter/second) obtained in the motion analysis laboratory
the parameters of gait analysis - cadence | through study completion, an average of 2 weeks (Change from Baseline parameters of gait analysis of the patients at 2 weeks.)
  cadence (number of steps/minute) obtained in the motion analysis laboratory
the parameters of gait analysis - single support time | through study completion, an average of 2 weeks (Change from Baseline parameters of gait analysis of the patients at 2 weeks.)
  single support time (second) obtained in the motion analysis laboratory
the parameters of gait analysis - double support time | through study completion, an average of 2 weeks (Change from Baseline parameters of gait analysis of the patients at 2 weeks.)
  double support time (second) obtained in the motion analysis laboratory
the parameters of gait analysis - contralateral foot contact time | through study completion, an average of 2 weeks (Change from Baseline parameters of gait analysis of the patients at 2 weeks.)
  contralateral foot contact time (second) obtained in the motion analysis laboratory
the parameters of gait analysis - step time | through study completion, an average of 2 weeks (Change from Baseline parameters of gait analysis of the patients at 2 weeks.)
  step time (second) obtained in the motion analysis laboratory
the parameters of gait analysis - step speed | through study completion, an average of 2 weeks (Change from Baseline parameters of gait analysis of the patients at 2 weeks.)
  step speed (centimeter/second)) obtained in the motion analysis laboratory
Walking Index for SCI - II (WISCI-II) Scale | through study completion, an average of 2 weeks (Change from Baseline WISCI II scale scores of the patients at 2 weeks.)
  Walking Index for SCI - II (WISCI-II) Scale (WISCI -II is a scale to assess the amount of physical assistance needed as well as device reuired for walking ( The development of this assessment index required a rank ordering along a dimension of impairment, from the level of most severe impairment (0) to least severe impairment (20) based on the use of devices, braces and physical assistance of one or more persons. The order of the levels suggests each successive level is a less impaired level than the former)
10-meter Gait Test | through study completion, an average of 2 weeks (Change from Baseline 10 meter gait test scores of the patients at 2 weeks.)
  10-meter Gait Test (This test is used to assess walking speed in meters per second over a short duration

CONTACTS AND LOCATIONS:
Overall Officials: SERDAR KESİKBURUN, MD, Study Director — The Scientific and Technological Research Council of Turkey; AYÇA URAN ŞAN, Principal Investigator — The Scientific and Technological Research Council of Turkey

IPD SHARING:
Plan to Share IPD: No